CLINICAL TRIAL: NCT06045325
Title: Assessment of Measurement Variability Across Automated Biometry Devices
Status: Completed | Type: Observational
Sponsor: Berkeley Eye Center (Other)
Responsible Party: Sponsor
Other Study IDs: BEC006
Record Dates: First submitted 2023-09-14; First posted 2023-09-21 (Actual); Results first posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Myopia
Keywords: -1.00 Diopter Spherical Equivalent
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Myopic -1.00D: Myopic patients with a diopter of at least -1.00
  Interventions: Diagnostic Test: Orbscan II; Diagnostic Test: IOL Master 700; Diagnostic Test: IOL Master 500; Diagnostic Test: Atlas 9000; Diagnostic Test: Lenstar 900; Diagnostic Test: Pentacam; Diagnostic Test: iTrace; Diagnostic Test: Argos; Diagnostic Test: Manual caliper measurement

INTERVENTIONS:
Diagnostic Test: Orbscan II — Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
Diagnostic Test: IOL Master 700 — Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
Diagnostic Test: IOL Master 500 — Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
Diagnostic Test: Atlas 9000 — Diagnostic assessment to measure white-to-white.
Diagnostic Test: Lenstar 900 — Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
Diagnostic Test: Pentacam — Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
Diagnostic Test: iTrace — Diagnostic assessment to measure white-to-white and corneal thickness.
Diagnostic Test: Argos — Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
Diagnostic Test: Manual caliper measurement — Manual diagnostic assessment to measure white-to-white.

SUMMARY:
This is a non-interventional prospective, comparative study of white-to-white, corneal thickness, and anterior chamber depth measurements as taken on the Orbscan II compared to the IOL Master 700 (Zeiss), IOL Master 500 (Zeiss), Atlas 9000 (Zeiss), Lenstar 900 (Haag-Streit), Argos (Alcon), iTrace (Tracey), Pentacam (Oculus), and manual calipers.

DETAILED DESCRIPTION:
This is a non-interventional prospective, single center, bilateral, comparative study of white-to-white, corneal thickness, and anterior chamber depth measurements as taken on the Orbscan II compared to the IOL Master 700 (Zeiss), IOL Master 500 (Zeiss), Atlas 9000 (Zeiss), Lenstar 900 (Haag-Streit), Argos (Alcon), iTrace (Tracey), Pentacam (Oculus), and manual calipers. Additional biometric devices or external photography may be included as well.

ELIGIBILITY:
Inclusion Criteria:

1. Adults ages 18-50 years of age with healthy eyes and no prior ocular surgery
2. At least -1.00 of myopia (spherical equivalent)
3. Able to comprehend and willing to sign informed consent and consent and complete all required testing procedures
4. Clear intraocular media

Exclusion Criteria:

1. Any corneal abnormality, other than regular corneal astigmatism (as determined by pre-operative testing) that in the opinion of the investigator would confound the outcome(s) of the study
2. History of or current retinal conditions or predisposition to retinal conditions
3. Amblyopia or strabismus in either eye
4. History of or current anterior or posterior segment inflammation of any etiology
5. Any form of neovascularization on or within the eye
6. Glaucoma (uncontrolled or controlled with medication)
7. Optic nerve atrophy
8. Subjects with diagnosed degenerative eye disorders
9. Subjects who have an acute or chronic disease or illness that would confound the results of this investigation in the opinion of the principal investigator (e.g. connective tissue disease, immunocompromised, clinically significant atopic disease, etc.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Myopic patients with a spherical equivalent of at least -1.00D with healthy eyes and no prior eye surgery.
Sampling Method: Non-Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2023-07-25 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morgan Micheletti, MD, Principal Investigator — Berkeley Eye Center
Locations (1):
- Berkeley Eye Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: eyes
Period: Overall Study
Arm/Group | Myopic -1.00D
Started | 204; 408 eyes
Completed | 204; 408 eyes
Not Completed | 0; 0 eyes

BASELINE CHARACTERISTICS:
Units Other Than Participants: eyes
Groups:
- Myopic -1.00D: Myopic patients with a diopter of at least -1.00. All patients will receive scans with each device.
  Orbscan II: Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
  IOL Master 700: Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
  IOL Master 500: Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
  Atlas 9000: Diagnostic assessment to measure white-to-white.
  Lenstar 900: Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
  Pentacam: Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
  iTrace: Diagnostic assessment to measure white-to-white and corneal thickness.
  Argos: Diagnostic assessment to measure anterior chamber depth, white-to-white, and corneal thickness.
  Manual caliper measurement: Manual diagnostic assessment to measure white-to-white.
Arm/Group | Myopic -1.00D
Number analyzed (Participants) | 204
Number analyzed (eyes) | 408
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 204
  >=65 years | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Not disclosed | 204
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0

OUTCOME MEASURES:

1. Primary Outcome: The Correlation of White-to-white Measurements Between Biometric Devices.
Description: The determination of the degree of correlation of white-to-white measurements between various biometric devices and the Orbscan II.
Time Frame: Day of visit
Measure: Number (95% Confidence Interval); unit: Pearson correlation r
Units Other Than Participants: eyes
Groups:
- Argos: Argos biometer
- Atlas 9000: Atlas 9000 biometer
- Manual Caliper: Manual Caliper
- IOLMaster 500: IOLMaster 500 biometer
- IOLMaster 700: IOLMaster 700 biometer
- iTrace: iTrace device
- Lenstar LS900: Lenstar LS900 biometer
- Pentacam AXL Wave: Pentacam AXL Wave device
- Pentacam HR: Pentacam HR device
Arm/Group | Argos | Atlas 9000 | Manual Caliper | IOLMaster 500 | IOLMaster 700 | iTrace | Lenstar LS900 | Pentacam AXL Wave | Pentacam HR
Number analyzed (Participants) | 204 | 204 | 204 | 204 | 204 | 204 | 204 | 161 | 204
Number analyzed (eyes) | 408 | 408 | 408 | 408 | 408 | 408 | 408 | 322 | 408
Pearson correlation r | 0.89 [0.87 to 0.91] | 0.65 [0.59 to 0.71] | 0.53 [0.46 to 0.60] | 0.60 [0.54 to 0.66] | 0.82 [0.78 to 0.85] | 0.78 [0.74 to 0.82] | 0.87 [0.84 to 0.89] | 0.84 [0.81 to 0.87] | 0.84 [0.81 to 0.87]

2. Primary Outcome: The Correlation of Anterior Chamber Depth Measurements Between Biometric Devices.
Description: The determination of the degree of correlation of anterior chamber depth measurements between various biometric devices and the Orbscan II.
Time Frame: Day of visit
Measure: Number (95% Confidence Interval); unit: Pearson correlation r
Units Other Than Participants: eyes
Arm/Group | Argos | IOLMaster 500 | IOLMaster 700 | Lenstar LS900 | Pentacam AXL Wave | Pentacam HR
Number analyzed (Participants) | 204 | 204 | 204 | 204 | 161 | 204
Number analyzed (eyes) | 408 | 408 | 408 | 408 | 322 | 408
Pearson correlation r | 0.91 [0.90 to 0.93] | 0.39 [0.31 to 0.47] | 0.33 [0.24 to 0.41] | 0.41 [0.33 to 0.49] | 0.95 [0.94 to 0.96] | 0.96 [0.96 to 0.97]

3. Primary Outcome: The Correlation of Corneal Thickness Measurements Between Biometric Devices.
Description: The determination of the degree of correlation of corneal thickness measurements between various biometric devices and the Orbscan II.
Time Frame: Day of visit
Population: Note that the iTrace, IOLMaster 500, Atlas 9000, and manual caliper did not measure central corneal thickness, so no central corneal thickness data were collected from these devices.
Measure: Number (95% Confidence Interval); unit: Pearson correlation r
Units Other Than Participants: eyes
Arm/Group | Argos | IOLMaster 700 | Lenstar LS900 | Pentacam AXL Wave | Pentacam HR
Number analyzed (Participants) | 204 | 204 | 204 | 161 | 204
Number analyzed (eyes) | 408 | 408 | 408 | 322 | 408
Pearson correlation r | 0.82 [0.78 to 0.85] | 0.80 [0.76 to 0.83] | 0.68 [0.63 to 0.73] | 0.68 [0.62 to 0.73] | 0.73 [0.68 to 0.77]

ADVERSE EVENTS:
Time Frame: Day of visit
Groups:
- Orbscan II: Orbscan II device
Arm/Group | Argos | Atlas 9000 | Manual Caliper | IOLMaster 500 | IOLMaster 700 | iTrace | Lenstar LS900 | Pentacam AXL Wave | Pentacam HR | Orbscan II
All-Cause Mortality (participants affected / at risk) | 0/204 | 0/204 | 0/204 | 0/204 | 0/204 | 0/204 | 0/204 | 0/161 | 0/204 | 0/204
Serious Adverse Events (participants affected / at risk) | 0/204 | 0/204 | 0/204 | 0/204 | 0/204 | 0/204 | 0/204 | 0/161 | 0/204 | 0/204
Other Adverse Events (participants affected / at risk) | 0/204 | 0/204 | 0/204 | 0/204 | 0/204 | 0/204 | 0/204 | 0/161 | 0/204 | 0/204

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT06045325/Prot_SAP_000.pdf